CLINICAL TRIAL: NCT05321381
Title: Thriving Together: Supporting Resilience in the Healthcare Workforce
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IRB00319396
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Emotional Distress; Burn Out; Anxiety
Keywords: Resilience; Well-being; Burnout; Health Care Worker; Peer Support
MeSH Terms: conditions — Burnout, Psychological; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Complete stepped-wedge cluster randomized design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RISE Early (Active Comparator): RISE peer support program available early, launched study year 1
  Interventions: Other: Resilience In Stressful Events (RISE) peer support team
- RISE Late (Active Comparator): RISE peer support program available later, launched study year 2
  Interventions: Other: Resilience In Stressful Events (RISE) peer support team

INTERVENTIONS:
Other: Resilience In Stressful Events (RISE) peer support team — Availability of peer support team to health care workers who experience stressful work-related events or situations

SUMMARY:
Health care workers (HCW) face distressing work related situations that pose a threat to the HCW's resilience and well-being. Hospital-based peer support programs can improve HCW well-being, but there are few programs and little data for settings outside of hospitals. The program would adapt, implement, and evaluate an evidence-informed peer support program (RISE) in ambulatory practices, rural hospitals, Federally Qualified Health Centers (FQHC), and community based organizations (CBOs). The hypothesis is that the availability of peer support will improve the culture of well-being, and the resilience and well-being of HCW in participating organizations. The research has the potential to improve the quality of life of HCW and the quality of care available to diverse organizations and the populations the HCW serve.

DETAILED DESCRIPTION:
Health care workers (HCW) face distressing work related situations that pose a threat to the HCW's resilience and well-being. Hospital-based peer support programs can improve HCW well-being, but there are few programs and little data for settings outside of hospitals. The program would adapt and implement an evidence-informed peer support program ((Resilience in Stressful Events = RISE) in ambulatory practices, rural hospitals, Federally Qualified Health Centers (FQHC), and community based organizations (CBOs). The hypothesis is that the availability of peer support will improve the culture of well-being, and the resilience and well-being of HCW in participating organizations.

The objectives are to:

1. Adapt and implement the RISE hospital peer support model in other health care contexts where HCW experience distressing events in the HCW's work.
2. Adapt and implement the Mental Emotional and Spiritual Help (MESH) collaborative model to provide a coordinated continuum of HCW support programs.
3. Adapt and implement a curriculum targeted at supporting organizational leaders during times of crisis which focuses on communication skills and understanding of fundamental psychological responses to stress.
4. Evaluate the program's effect on the culture of wellbeing, and the resilience and well-being of HCW in participating organizations.

The design of the study is a mixed-methods evaluation of the implementation of training and organizational structures to support HCW at different types of healthcare organizations (45 John Hopkins Community Physicians (JHCP) outpatient primary care clinics, 3 rural hospitals, 3 Federally Qualified Health Centers, and 3 community-based social service organizations - for a total 54 practice sites).

Based on the training, participating organizations will develop the organizations' own volunteer-based team to provide confidential, timely, peer support for HCW who encounter stressful, patient-related events. The RISE team is available on-call 24/7 to respond to calls and provide in person or virtual psychological first aid sessions.

The primary evaluation will be based on the differences between anonymous pre and post implementation surveys of random samples of HCW across sites. In the cluster randomized design, each of the 54 practice sites is considered a cluster. Half of the sites will be randomized to receive a team of trained RISE peer supporters launching in Year1Quarter3. The other half will receive this services launching Year2Quarter3.

The baseline survey will be in Year1Quarter2, the step 1 survey will be in Year2Qquarter2, and the step 2 survey will be Year3Quarter2. A random sample of 352 HCW will be surveyed at each time point. Focus groups will be conducted during the intervention with 120 HCW to inform quality improvement, and with 160 HCW across types of organization to coincide with the step 1 and step 2 surveys, to ask about the uptake of peer support services.

Survey data collection will be anonymous via a secure online platform. Focus groups will be conducted virtually using Zoom. HCWs will be compensated to complete surveys and participate in focus groups.

Analysis: The investigators will aim to detect a change of 0.2-0.3 standard deviation (SD) units on a given scale score, from before until after implementation, between the different steps. The investigators assume an intra-cluster (within site) correlation (ICC) of 0.3 SD. To detect an effect size of 0.3 on a measure of anxiety (GAD-7) for independent survey samples pre- and post-intervention step, with a two-tailed alpha=0.05 and power=80%, the investigators would need a total of 1056 HCW responses (352 at each of 3 survey timepoints) using a two-sided Wald Z-Test.

ELIGIBILITY:
Inclusion Criteria:

* Health care worker employed at participating implementation health care site/organization

Exclusion Criteria:

* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1362 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Generalized Anxiety Disorder-7 scale (GAD-7) score | Baseline, 1 and 2 years
  Score on 7-item scale to measure anxiety

SECONDARY OUTCOMES:
Change in Adult PROMIS Short Form v.1.0 Sleep Disturbance 4a score | Baseline, 1 and 2 years
  Score on single item to measure sleep disturbance : Adult Patient Reported Outcome Measurement Information System (PROMIS) Short Form v.1.0 Sleep Disturbance 4a.
Change in Impact of Event Scale-Revised (IES-R) score | Baseline, 1 and 2 years
  Score on scale to measure post traumatic stress.
Change in Maslach Burnout Inventory 2-item (MBI-2) scale score | Baseline, 1 and 2 years
  Score on 2-item scale to measure worker burnout.
Change in Connor-Davidson Resilience Scale 2-item score | Baseline, 1 and 2 years
  Score on 2-item scale to measure resilience.
Change in Patient Health Questionnaire-2 (PHQ-2) score | Baseline, 1 and 2 years
  Score on 2-item scale to measure depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Albert W Wu, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Community Physicians, Baltimore, Maryland
  - UM Shore Regional Health, Chestertown, Maryland

IPD SHARING:
Plan to Share IPD: No